CLINICAL TRIAL: NCT01251874
Title: A Phase 1 Dose-Escalation Study of ABT-888 (Veliparib) in Combination With Carboplatin in HER2 Negative Metastatic Breast Cancer
Brief Title: Veliparib and Carboplatin in Treating Patients With HER2-Negative Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02552; NCI-2011-02552 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000688990; OSU 10080; 8609 (Other: Ohio State University Comprehensive Cancer Center); 8609 (Other: CTEP); P30CA016058 (NIH); U01CA076576 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Breast Carcinoma; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Specimen Handling; Carboplatin; alovudine; Magnetic Resonance Spectroscopy; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (veliparib, F 18 fluorothymidine, carboplatin) (Experimental): Patients receive carboplatin IV over 1 hour on day 1 and veliparib PO BID on days 1-7 or 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients may undergo fluorothymidine PET scan and peripheral blood cell and tumor tissue collection periodically for correlative studies.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Other: Fluorothymidine F-18; Procedure: Positron Emission Tomography; Drug: Veliparib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Fluorothymidine F-18 — Given FLT
  Other Names: 18F-FLT; 3'-Deoxy-3'-(18F) Fluorothymidine; 3'-deoxy-3'-[18F]fluorothymidine; ALOVUDINE F-18; Fluorothymidine F 18
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I trial studies the side effects and best dose of veliparib when given together with carboplatin and to see how well they work in treating patients with human epidermal growth factor 2 (HER2)-negative breast cancer that has spread to other parts of the body. Carboplatin kills cancer cells by damaging the deoxyribonucleic acid (DNA) that lets the cancer cell survive and reproduce. The body has proteins that try to repair the damaged DNA. Veliparib may prevent these proteins from repairing the DNA so that carboplatin may be able to kill more tumor cells. Giving veliparib with carboplatin may kill more tumor cells than carboplatin alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose of veliparib along with carboplatin on a 14-day and 21-day schedule in patients with Her2 negative metastatic breast cancer that are estrogen receptor (ER)/progesterone receptor(PR) negative or ER and/or PR positive with defects in Fanconi Anemia (FA) pathway repair genes.

II. To determine the safety and tolerability of combining veliparib on a 14-day and 21-day schedule with carboplatin in this patient population.

III. To determine the preliminary efficacy of this combination in this patient population.

SECONDARY OBJECTIVES:

I. To determine the pharmacodynamic endpoints of poly(ADP-ribose) polymerase (PARP) inhibition in the tumor by using, A) 3'-[F-18]fluoro-3'-deoxythymidine positron emission tomography (FLT-PET) of the target lesions, B) circulating tumor cells to detect the induction of the histone variant gamma H2AX, and C) peripheral blood mononuclear cells to assess poly ADP-Ribose (PAR) levels.

II. To determine biomarkers in the primary tumor that may predict antitumor responses to PARP inhibition such as breast cancer 1/2, early onset (BRCA)1/2 protein, Fanconi anemia, complementation group D2 (FANCD2) nuclear foci formation and expression of micro-ribonucleic acid (RNA) 155 (miR 155).

OUTLINE: This is a dose-escalation study of veliparib.

Patients receive carboplatin intravenously (IV) over 1 hour on day 1 and veliparib orally (PO) twice daily (BID) on days 1-7 or 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Additionally, patients also undergo collection of blood sample, positron emission tomography (PET)/computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed up for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically proven metastatic or locally advanced inoperable breast cancer that fulfills one of the following two criteria:

  * Triple-negative breast cancer
  * ER and/or PR positive, HER2 negative if their tumors have been shown to be deficient for the FA pathway, based on FA triple stain immunofluorescence (FATSI) screening
  * HER negative with a known germline BRCA1/2 mutation

    * Patients with ER- and/or PR-positive breast cancer will be consented to have their existing, or to be obtained, paraffin-embedded tumor tissue screened for FA deficiency
* No more than 3 prior chemotherapy regimens for metastatic disease will be allowed; any number of prior hormone therapies will be allowed; however, at least 4 weeks should have elapsed since prior chemotherapy (6 weeks for mitomycin C and nitrosoureas and 2 weeks for hormone therapy) or radiation therapy (2 weeks for limited field palliative radiation to the bone)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Patients with treated brain metastases and life expectancy of greater than 3 months
* Patients with known Gilbert syndrome with abnormal unconjugated bilirubin will be eligible
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic acid transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* No prior therapy with veliparib for metastatic disease will be allowed
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients must be able to swallow pills

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to veliparib or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with veliparib
* Known human immunodeficiency virus (HIV)-infected patients on protease inhibitors are ineligible; HIV-infected patients with adequate cluster of differentiation (CD)4 counts (> 500) and not on protease inhibitors are eligible
* Patients with active seizure or a history of seizures are not eligible
* Patients with uncontrolled central nervous system (CNS) metastasis are not eligible; patients with CNS metastases must be stable after therapy for > 3 months and off steroid treatment prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events to measure the safety and tolerability of this treatment combination | Up to 12 weeks post-treatment
  Number and severity of toxicity incidents will be tabulated. Non-hematologic toxicities will be evaluated via the ordinal Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir and percent change from baseline values) as well as categorization via CTCAE standard toxicity grading. Frequency distributions and other descriptive measures will form the basis of the analysis of these variables.

SECONDARY OUTCOMES:
Clinical response (complete and partial response as well as stable and progressive disease) | Up to 12 weeks post-treatment
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease. Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors guideline (version 1.1).

OTHER OUTCOMES:
PARP-1 activity | Up to 5 years
  Analysis will be descriptive and exploratory in nature. Potential relationships and differences will be explored using graphical analyses and quantitative summaries of this marker.
Thymidine kinase uptake on 3'-[F-18]fluoro-3'-deoxythymidine positron emission tomography (FLT-PET) scans | Up to 18 weeks (after course 3)
  Analysis will be descriptive and exploratory in nature. Potential relationships and differences will be explored using graphical analyses and quantitative summaries of this marker.
Circulating tumor cell markers | Up to 5 years
  Analysis will be descriptive and exploratory in nature. Potential relationships and differences will be explored using graphical analyses and quantitative summaries of this marker.

CONTACTS AND LOCATIONS:
Overall Officials: Kai C Johnson, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio